CLINICAL TRIAL: NCT03987464
Title: Platform-Based Mild Cognitive Impairment (MCI) Trial to Address Maladaptive Behaviors
Brief Title: Platform-based Mild Cognitive Impairment (MCI) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allison Gibson (Other)
Responsible Party: Sponsor-Investigator, Allison Gibson, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 44035
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Mild Cognitive Impairment
Keywords: Alzheimer's Disease; maladaptive; behavior
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with MCI (Experimental): Participants diagnosed with mild cognitive impairment (MCI) and their study partners
  Interventions: Behavioral: Planning for the Future; Behavioral: Enhanced Medical Engagement; Behavioral: Confidence Building and Social Engagement; Behavioral: Physical Intervention; Behavioral: Medical Adherence

INTERVENTIONS:
Behavioral: Planning for the Future — This intervention will include attending an advance directives meeting, a living arrangements workshop, and a psychosocial education training workshop.
Behavioral: Enhanced Medical Engagement — This intervention includes creating a health portfolio, health record access training, and a medical engagement workshop
Behavioral: Confidence Building and Social Engagement — This intervention includes mindfulness training, a pre-experience training techniques workshop and a memory strategies class.
Behavioral: Physical Intervention — This intervention includes physical/occupational therapy (PT/OT), a home safety assessment, and an independent exercise program.
Behavioral: Medical Adherence — This intervention includes using automated pillboxes to ensure medication compliance, optimizing appropriate medication use through review, and engaging with memory medications via class.

SUMMARY:
The process of receiving a diagnosis of mild cognitive impairment (MCI) is recognized to induce behavioral responses that can be either adaptive or maladaptive. Five specific areas of concern have been identified, including: 1) failure to plan for future decline, decreased compliance and interaction with medical care providers, 3) decreased confidence and reduced social engagement, 4) increased physical limitations and 5) decreased medication compliance. In this pilot study, participants with MCI and their study partners will participate in behavioral interventions (primarily training workshops and classes) targeting each of these five areas of potential maladaptive behaviors.

DETAILED DESCRIPTION:
Following the approval of an application reviewed by the University's Institutional Review Board, the researcher will evaluate the intervention using a complimentary mixed methods approach. The study will consist of a single-site platform trial examining the intervention group. There are many benefits to using a platform trial approach. First, using a platform trial allows the 18 participants to explore different arms of the intervention. Second, the platform design will allow us to also determine the effects of the interventions on patient help-seeking and adherence behavior in real-world care is critical to estimates of cost-effectiveness. As one of the specific aims of this study is to determine user feedback about modifying behaviors from various interventions, as opposed to determining which intervention is most effective, a platform trial will accomplish this.

ELIGIBILITY:
Inclusion Criteria:

* current subjects of the University of Kentucky Alzheimer's Disease Center (ADC)
* meet consensus guidelines for mild cognitive impairment (MCI) developed by the Second International Working Group on MCI
* have been diagnosed within the last year
* able to provide informed consent
* have a study partner willing to participate

Exclusion Criteria:

* history of stroke
* significant neurological or psychiatric conditions
* brain injury
* residence in institutional setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy; general self-efficacy scale (GSES) | 9 months
  The general self-efficacy scale (GSES) is a ten-item scale. Scores range from 10-40, with higher scores indicating more self-efficacy.

SECONDARY OUTCOMES:
Readiness to complete advance directives (ACPES) | 9 months
  The readiness to complete advance directives is a 4-item scale. Scores range from 4-20, with higher scores indicating more readiness to complete advance directives.
Motivations Around Advance Care Planning (ADS) | 9 months
  The motivations around advance care planning is a 9-item scale. Scores range from 9-45, with higher scores indicating motivational influences for advance care planning decisions
Long Term Care Planning Behavior Scale (LTCP), planning subscale | 9 months
  The considered future living arrangement is a 3-item subscale. Scores range from 3-15, with higher scores indicating higher knowledge about future living arrangement options.
Long-Term Supports and Services (LTSS) | 9 months
  The long-term supports and services is an 11-item scale. Scores range from 0-11, with higher scores indicating being more open to long-term support and service options.
World Health Organization Quality-of-Life (WHOQOL), Brief - Psychological and Social Relationship subscale | 9 months
  WHOQOL psychological and social relationships is an 9-item subscale. Scores range from 9-25, with higher scores indicating a higher quality-of-life.
MCI Test of Knowledge (MCI-ToK) | 9 months
  The long-term supports and services is an 5-item scale. Scores range from 0-5, with higher scores indicating a higher level of knowledge about MCI.
Long Term Care Planning Behavior Scale (LTCP), health subscale | 9 months
  The LTCP health subscale is 3-items. Scores range from 0-12, with higher scores indicate willingness to follow directions about healthcare supports and services.
Technophilia Scale, Technology for health subscale (TTfH) | 9 months
  The Technophilia Scale-Technology for health subscale is 2-items. Scores range from 2-10, with higher scores indicate a higher rate of use of technology for one's health.
Technophilia Scale, Comfort with technology subscale (TCwT) | 9 months
  The Technophilia Scale-Comfort with technology is a 4-item scale. Scores range from 4-20, with higher scores indicate a higher rate of perceived comfort with using technology.
Technophilia Scale, Use of technology subscale (TUoT) | 9 months
  The Technophilia Scale-Use of technology is 3-items. Scores range from 3-15, with higher scores indicating more frequent use of technology.
Patient communication pattern scale (PCPS) | 9 months
  The PCPS is a 14-item scale. Scores range from 14-84, with higher scores indicating higher rates of communication with healthcare professionals.
Comfort engaging medical professionals (CEMP) | 9 months
  The CEMP is a 4-item scale. Scores range from 4-20, with higher scores indicating more more comfort with engagement with medical care.
Mindfulness Attention Awareness Scale (MAAS) | 9 months
  The MAAS is a 6-item scale. Scores range from 6-90, with higher scores indicating higher awareness of daily thoughts and tasks.
Mindfulness Adherence Questionnaire (MAQ) | 9 months
  The MAAS is a 4-item scale. Scores range from 0-20, with higher scores indicating higher rates of adherence to the practice of mindfulness.
CHAMPS Physical Activity Questionnaire for Older Adults (CHAMPS), Social engagement subscale. | one month
  The CHAMPS's social engagement is a 5-item subscale. Scores range from 0-30, with higher scores indicating higher rates of social engagement.
Social Interaction Anxiety Scale (SIAS) | 9 months
  The SIAS is a 6-item scale. Scores range from 0-12, with higher scores indicating higher levels of social interaction anxiety.
Crowne-Marlowe Social Desirability (CMSDS) | 9 months
  The CMSDS includes 2-items. Scores range from 0-2, with lower scores indicating higher levels of social desirability.
Memory Situation Questionnaire (MSQ; adapted) | 9 months
  The MSQ includes 5-item scale. Scores range from 0-5, with higher scores indicating higher knowledge of memory strategies.
Sickness Impact Profile (SIP) - subscales including body care and movement, mobility, and home management | 9 months
  The SIP subscales include 6-items. Scores range from 0-6, with higher scores indicating higher impact of illness.
CHAMPS Physical Activity Questionnaire for Older Adults (CHAMPS), Physical activity subscale | 9 months
  The CHAMPS's social engagement is a 7-item subscale. Scores range from 0-35, with higher scores indicating higher rates of physical activity.
Long Term Care Planning Behavior Scale (LTCP), home modifications item | 9 months
  This is 1 item on home modifications. Scores range from 0-1, with "0" representing no home modifications to prepare for the future and "1" indicating changes home modifications made to prepare for the future.
Short Falls Efficacy Scale (Short FES-I) | 9 months
  The SIP subscale includes 7-items. Scores range from 0-28, with higher scores indicating higher concern for falls.
36-Item Short Form Survey (SF-36) - physical functioning, pain, energy/fatigue, subscales | 9 months
  These subscales include 16-items. Scores range from 16-61, with lower scores indicating higher limitations to physical functioning.
Activity | 9 months
  Uniaxial accelerometer (MTI) measured activity counts
Medication Adherence (MA-MCI) | 9 months
  The Medication Adherence scale includes 3-items for the MCI subjects. Scores range from 3-15, with lower scores indicating higher medication adherence.
Medication Adherence (MA-SP) | 9 months
  The Medication Adherence scale includes 3-items and is for the subjects that are study partners to the participant diagnosed with MCI. Scores range from 3-15, with lower scores indicating higher medication adherence.
Concerns about Memory Medications (CaMM) | 9 months
  This is 1 item. Scores range from 0-1, with "0" not adhering to medication and "1" is adhering to medication.
Motivations around Memory Medications (MMM) | 9 months
  The Motivations around Memory Medications scale includes 4-items. Scores range from 5-20, which measures attitudes around memory medications. Higher score indicates more positive attitudes about taking memory medications.
MCI Medication Test of Knowledge (MCI-MToK) | 9 months
  The MCI Medication Test of Knowledge scale includes 4-items. Scores range from 0-4 where a higher score indicates a higher level of medication knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Gibson, PhD, MSW, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No